CLINICAL TRIAL: NCT01918163
Title: Anti-oxidative Influence From Pomegranate Tablets on Male Sperm Quality in Couples Undergo Infertility Treatments Due to Male Infertility.
Acronym: Pomegranate
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 0059-13HYMC
Record Dates: First submitted 2013-07-14; First posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-07

CONDITIONS: Male Infertility With Severe Oligo-terato-asteno-spermia
Keywords: pomegranate pills, male infertility, pregnancy rate, semen analysis, ROS, oxidative stress
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Pills (No Intervention): Patients in this group will not receive Pomegranate pills.
- Pomegranate pills (Active Comparator): The reccruited patient will receive pomegranate pills every day for 12 weeks. The control group will not be exposed for the pills.
  Interventions: Dietary Supplement: Pomegranate pills

INTERVENTIONS:
Dietary Supplement: Pomegranate pills
  Arms: Pomegranate pills

SUMMARY:
Some animal studies revealed that the pomegranate juice may improve sperm quality in terms of concentration, motility and morphology, as well as in fertilization rate.

Minor data is available regarding the influence on male sperm.

DETAILED DESCRIPTION:
Pomegranate contains a high concentration of vitamins ( C, B1, B2, B3, B5), potassium, Magnesium , Zinc and is a good source for polyphenols .Polyphenols molecules have been found to possess antioxidant properties and may effects the expression of different genes . Recent studies indicate that among foods that contain polyphenols, juice extracted from the pomegranate has the highest concentration of measurable polyphenols . Pomegranates have shown inhibitory effect on NF-κB and the MAP kinases JNK and ERK, which are critical steps in the cascade of events leading to inflammatory response. The NF- κB pathway is activated in response to bacterial infection and initiates the inflammatory cascade, which may explain the protective effect of Pomegranates on bacterial infections.

ELIGIBILITY:
Inclusion Criteria:

* TMC of less than 5 million spermatogonia in native sperm and morphology less than 4% by Kruger criteria.

Exclusion Criteria:

* sensitivity to Pomegranate

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
pregnancy | 24 month

SECONDARY OUTCOMES:
ROS (reactive oxidative stress )and Interleukins level in semen fluid | 12 weeks
  The unit for measure the ROS are Micromolar epicatechin equivalent

CONTACTS AND LOCATIONS:
Overall Officials: Einat Shalom-Paz, MD, Principal Investigator — Hillel Yaffe Medical center, IVF unit, Hadera, Israel
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel